CLINICAL TRIAL: NCT05973019
Title: Repetitive Transcranial Magnetic Stimulation Improves Functional Performance in Spinocerebellar Ataxia
Brief Title: rTMS Improves Functions in Spinocerebellar Ataxia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Principal Investigator, Sen-yung Liu, Chief Medical Officer, Changhua Christian Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 230425
Record Dates: First submitted 2023-07-25; First posted 2023-08-02 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Transcranial Magnetic Stimulation; Spinocerebellar Ataxias
Keywords: rTMS; SCA
MeSH Terms: conditions — Spinocerebellar Ataxias | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: All subjects receive 12 times rTMS intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- rTMS with 10 Hz (Experimental): 6 times/per week for 2 weeks, total 12 times rTMS.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — 6 times/per week for 2 weeks, total 12 times rTMS with 10 Hz.

SUMMARY:
Spinocerebellar ataxia (SCA) is a group of inherited brain disorders. SCA often result in poor limb coordination. This study aims to discover the effects of repeated transcranial magnetic stimulation (rTMS) on balance & gait in SCA. The hypothesis of this study is that rTMS might improve SCA limb functional performance.

DETAILED DESCRIPTION:
rTMS has been shown that improves walking speed and balance performance, however, the optimal treatment protocols have not been approved. Past studies used different frequencies 1 Hz, 5 Hz and 10 Hz to improve functional performance. The results might be affected by the types of SCA. In this study, we will focus on the SCA type 3 to assess the effects on high frequency (10 Hz) of rTMS intervention.

ELIGIBILITY:
Inclusion Criteria:

* SCA type 3
* independently walk with/without an assistive device
* SARA greater than 3

Exclusion Criteria:

* Epilepsy history
* Unstable blood pressure
* Brain Trauma
* Alcoholism, drug abuse, antipsychotics drug use
* Metallic hardware (e.g. - cochlear implants, brain stimulators or electrodes, aneurysm clips) anywhere in head.
* Dementia, depression

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Changes of International Cooperative Ataxia Rating Scale | Baseline (T0), 6 days after first rTMS intervention (T1), 12 days after first rTMS intervention (T2),
  International Cooperative Ataxia Rating Scale (ICARS): quantify the level of impairment as a result of ataxia as related to hereditary ataxias. Disorders rated as subscales within the ICARS are: Postural and gait disturbances, Limb Ataxia, Dysarthria, and Oculomotor disorders.It translates the symptomatology of cerebellar ataxia into a scoring system out of 100.
Changes of SARA | Baseline (T0), 6 days after first rTMS intervention (T1), 12 days after first rTMS intervention (T2),
  Scale for the Assessment and Rating of Ataxia (SARA): a tool for assessing ataxia. It has eight categories with accumulative score ranging from 0 (no ataxia) to 40 (most severe ataxia).
Changes of Berg Balance Scale | Baseline (T0), 6 days after first rTMS intervention (T1), 12 days after first rTMS intervention (T2),
  Berg Balance Scale (BBS): a widely used assessment to determine a person's balance abilities. The test contains 14 simple tasks, scoring ranges from 0 to 56. The lower your score, the more at risk you are for losing your balance. The entire process takes about 20 minutes to complete.
Changes of Timed up and go | Baseline (T0), 6 days after first rTMS intervention (T1), 12 days after first rTMS intervention (T2),
  Timed up and go (TUG): Patients wear their regular footwear and can use a walking aid, if needed. Begin by having the patient sit back in a standard arm chair and identify a line 3 meters, or 10 feet away, on the floor.
Changes of Center of pressure trajectory | Baseline (T0), 6 days after first rTMS intervention (T1), 12 days after first rTMS intervention (T2),
  Center of pressure (COP): he trajectory of the COP, commonly known as a stabilogram, during static balance is frequently used to measure postural control. When standing still on a force platform, the COP is thought to be an indicator of the motor mechanisms involved in maintaining balance with opened-eyes or closed-eyes. Two trials for each condition were performed within 5 minutes.
Changes of Kinematic of Gait | Baseline (T0), 6 days after first rTMS intervention (T1), 12 days after first rTMS intervention (T2),
  The joint angles of hip, knee, ankle are collected during walking in a 10 meters walkway.
Changes of Electromyography of Gait | Baseline (T0), 6 days after first rTMS intervention (T1), 12 days after first rTMS intervention (T2),
  A wireless surface Electromyography (EMG) is used to collect lower extremities muscle activation signals during walking in a walkway.

SECONDARY OUTCOMES:
Concentration of Neurofilament | Baseline (T0), 12 days after first rTMS intervention (T2)
  neurofilament proteins is the biomarkers of axonal damage in diseases affecting the central nervous system
Changes of Mini-mental state examination | Baseline (T0)
  The mini-mental state examination (MMSE) is a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment. A score of 25 or higher is classed as normal. If the score is below 24, the result is usually considered to be abnormal, indicating possible cognitive impairment. In this study, it is used to rule out subjects who might have dementia.

CONTACTS AND LOCATIONS:
Overall Officials: Sen Yung Liu, MD, Principal Investigator — Changhua Christian Hospital
Locations (1):
- Changhua christian hospital, Changhua, Taiwan